CLINICAL TRIAL: NCT01055678
Title: Pilot Study to Characterize the HRHV Axis in the Microenvironment of Breast Cancers
Brief Title: To Evaluate the Characteristics of a Breast Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI left Duke
Sponsor: Mark Dewhirst (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mark Dewhirst, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00020382; R01CA040355 (NIH)
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; ductal breast carcinoma in situ; breast cancer in situ; invasive carcinoma; invasive ductal carcinoma; invasive lobular carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Carcinoma, Lobular | interventions — Mastectomy, Simple

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Patients (Experimental): Single arm study analyzing tumor hypoxia after EF5 injection
  Interventions: Drug: EF5; Procedure: Partial or Total Mastectomy

INTERVENTIONS:
Drug: EF5 — An infusion of EF5, a fluorinated 2-nitroimidazole, will be administered using the recommended dose of 21mg/kg one day prior to surgical procedure.
Procedure: Partial or Total Mastectomy — A small tissue sample will be removed from the excised tissue and will be stored for later analysis.

SUMMARY:
The purpose of this pilot study is to determine the prevalence of markers of chronic and cycling hypoxia and reactive species stress (oxidative and nitrosative) in the breast cancer tumor microenvironment. The study is based around four cornerstone features of the pathologic microenvironment - Hypoxia, Reactive Species (reactive oxygen and nitrogen species), HIF-1 and VEGF, which we term the HRHV axis. Fifty breast cancer patients with planned surgical excision will be administered the hypoxia marker drug, EF5, 24-36 hr prior to surgical excision. EF5 is a non-therapeutic drug and provides no direct benefit to those patients enrolled in this pilot study. Tissues obtained intra-operatively will be snap frozen and subsequently analyzed for EF5 binding. Immunohistochemical analysis of a cohort of immunohistochemical and urine markers that depict the HRHV axis will be examined. The association of the markers with the presence of hypoxia, as determined by EF5 positivity, will be determined. Data from this pilot study will be used to establish the prevalence of markers of the HRHV axis in breast cancer. This information will be crucial for future human trials in which the HRHV axis is therapeutically targeted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage 0 - III invasive carcinoma of the breast
* Tumor size greater than 1-cm by radiological (mammogram/ultrasound or MRI) evaluation
* KPS status ≥ 70
* Bilirubin ≤ 1.5x normal
* Creatinine ≤ 1.8
* WBC > 3000/mm^3 and platelets > 100,000/mm^3

Exclusion Criteria:

* Pregnant or breast-feeding women
* Neoadjuvant chemo or hormonal therapy for existent breast malignancy
* Allergy to IV contrast dye
* History of grade III or IV peripheral neuropathy as defined by the NCI CTC
* Previous history of any malignancy treated with radiotherapy and/or chemohormonal therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To evaluate tumor characteristics | 2 years

SECONDARY OUTCOMES:
Intra and Interpatient correlations with tumor hypoxia | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Dewhirst, DVM, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Dewhirst MW, Cao Y, Moeller B. Cycling hypoxia and free radicals regulate angiogenesis and radiotherapy response. Nat Rev Cancer. 2008 Jun;8(6):425-37. doi: 10.1038/nrc2397. PMID 18500244
- [Background] Koch CJ, Hahn SM, Rockwell K Jr, Covey JM, McKenna WG, Evans SM. Pharmacokinetics of EF5 [2-(2-nitro-1-H-imidazol-1-yl)-N-(2,2,3,3,3-pentafluoropropyl) acetamide] in human patients: implications for hypoxia measurements in vivo by 2-nitroimidazoles. Cancer Chemother Pharmacol. 2001 Sep;48(3):177-87. doi: 10.1007/s002800100324. PMID 11592338